CLINICAL TRIAL: NCT04132713
Title: Study on Skin Microbiota of Hand Foot Syndrome
Brief Title: Study on Skin Microbiome of HFS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2019-09-12
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Microbiota
Keywords: skin microbiota; 16S rRNA gene; hand foot sysdom; breast cancer chemotherapy
MeSH Terms: interventions — Capecitabine; Tablets

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: 20 healthy volunteers were included in the healthy control group
- Disease group: 30 patients with advanced breast cancer developed hand-foot syndrome after capecitabine administration
  Interventions: Drug: Capecitabine 150Mg Oral Tablet

INTERVENTIONS:
Drug: Capecitabine 150Mg Oral Tablet — Advanced breast cancer patients with first-line medication
  Groups: Disease group

SUMMARY:
To skin microecology and breast cancer chemotherapy drug therapy as the breakthrough point, disease prevention and treatment of breast cancer in China, the important scientific problems in basic research, through in-depth study of skin micro ecological changes in advanced breast cancer chemotherapy and its regulatory mechanism, clear skin flora occurred after application of capecitabine and the influence and mechanism of the immune response;Finding markers for the treatment and prognosis of related diseases;Identify and isolate key strains and/or metabolites, and conduct intervention studies to reveal new mechanisms of skin microflora homeostasis and toxic and side effects of breast cancer chemotherapy.

DETAILED DESCRIPTION:
To skin microecology and breast cancer chemotherapy drug therapy as the breakthrough point, disease prevention and treatment of breast cancer in China, the important scientific problems in basic research, through in-depth study of skin micro ecological changes in advanced breast cancer chemotherapy and its regulatory mechanism, clear skin flora occurred after application of capecitabine and the influence and mechanism of the immune response;Finding markers for the treatment and prognosis of related diseases;Identify and isolate key strains and/or metabolites, and conduct intervention studies to reveal new mechanisms of skin microflora homeostasis and toxic and side effects of breast cancer chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* age: 18-65 years old
* advanced breast cancer patients
* healthy volunteers

Exclusion Criteria:

* previous skin disease history, or other skin disease activity at present
* various antibiotics, prebiotics, probiotics or lactic acid products used within three months;
* having a history of alcoholism for more than 2 years and smoking for years;
* pregnancy or lactation;
* have oral, respiratory and gastrointestinal diseases;
* other metabolic diseases, such as obesity, hypertension, diabetes, stones, and liver diseases;
* other autoimmune diseases, such as rheumatoid arthritis, ankylosing spondylitis, inflammatory bowel disease;
* history of gastrointestinal surgery;
* family genetic history, history of mental illness, etc.;
* the subject is participating in other research projects;
* other reasons are not considered suitable for continued clinical trials.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients were included according to the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Transcriptional changes in skin microbiota | baseline,1 day, 21 days,42 days,65 days,85 days,106 days,127 days
  The microbiota measured by 16S rRNA gene

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weese JS. The canine and feline skin microbiome in health and disease. Vet Dermatol. 2013 Feb;24(1):137-45.e31. doi: 10.1111/j.1365-3164.2012.01076.x. PMID 23331690
- [Background] Kong HH, Segre JA. Skin microbiome: looking back to move forward. J Invest Dermatol. 2012 Mar;132(3 Pt 2):933-9. doi: 10.1038/jid.2011.417. Epub 2011 Dec 22. PMID 22189793
- [Background] Roth RR, James WD. Microbiology of the skin: resident flora, ecology, infection. J Am Acad Dermatol. 1989 Mar;20(3):367-90. doi: 10.1016/s0190-9622(89)70048-7. PMID 2645319